CLINICAL TRIAL: NCT00687050
Title: MRT-based Pilot Study to Evaluate Peroral Supplemental Nutrition for Prevention of Cachexia in End-stage Renal Disease With and Without HIV Comorbidity
Brief Title: Peroral Supplemental Nutrition in End-stage Renal Disease With and Without HIV Comorbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Pfrimmer Nutricia GmbH, Erlangen , Germany (Industry)
Responsible Party: Dr. Rainer U. Pliquett, Goethe University Frankfurt am Main
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Goethe-Uni-FFM-328-07
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: End-Stage Renal Disease
Keywords: end-stage renal disease; chronic kidney disease
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): HIV-positive hemodialysis patients (as a high risk group for cachexia) will be given daily drinks of Renilon 7.5 (125 ml, 2 kcal/ml) as peroral supplemental nutrition on top to their recommended high-protein, high-caloric diet.
  Interventions: Dietary Supplement: peroral high-caloric supplemental nutrition
- 2 (No Intervention): Chronic hemodialysis patients randomized to no peroral supplemental nutrition
- 3 (Active Comparator): Chronic hemodialysis patients randomized to peroral supplemental nutrition.
  Interventions: Dietary Supplement: peroral supplemental nutrition

INTERVENTIONS:
Dietary Supplement: peroral high-caloric supplemental nutrition — HIV-positive hemodialysis patients will be given daily supplemental nutrition (125 ml, 2 kcal/ml) on top of recommended high-protein, high-caloric regular diet
  Other Names: Renilon 7.5 by Pfrimmer Nutricia
  Arms: 1
Dietary Supplement: peroral supplemental nutrition — Chronic hemodialysis patients will be given daily peroral supplemental nutrition (125 ml/d, 2 kcal/ml) on top of their recommended high-protein, high caloric diet
  Other Names: Renilon 7.5 by Pfrimmer-Nutricia
  Arms: 3

SUMMARY:
End-stage renal disease is often accompanied by malnutrition due to less appetite, metabolic changes or both. Human immunodeficiency virus-infection may exacerbate the state of malnutrition. In a pilot study, we recruit both HIV invected and non-infected patients on hemodialysis. Non-HIV patients will be randomized to peroral supplemental nutrition or no peroral supplemental nutrition. All HIV patients will receive peroral supplemental nutrition. The nutritional state will be determined in magnet resonance tomography at the start and at the end of the study (muscle diameter of triceps m.) and with laboratory parameters (plasma albumin and others). The hypothesis is that supplemental peroral nutrition (a total 250 kcal per day) will stop loss of muscle mass in end-stage renal disease patients (compared to their counterparts without supplemental peroral nutrition) as well as in the high risk group of HIV patients. This pilot study may lead to larger randomized clinical trials and, may affect dietary recommendations.

DETAILED DESCRIPTION:
In end-stage renal disease (ESRD), cachexia is a common finding. Metabolic changes, malnutrition, or both appear to be the underlying problems. In fact, lean body mass per body weight better predicts prognosis than creatinin based models (NDT, 2004.19:1182). In addition, comorbidity such as HIV infection may exacerbate cachexia found in ESRD. Whether or not daily supplemental, high-caloric nutrition in ESRD corrects a catabolic state in ESRD is unclear.

Hypothesis to be tested:

Daily supplemental high-caloric nutrition beneficially affects cytokine stimulation (TNF alpha, IL 1beta, IL 6, CrP) and nutritional state (cross sectional area of triceps m. in mid-humerus position (MRT), plasma albumin) in in HIV-positive hemodialysis patients and in chronic hemodialysis patients compared to chronic hemodialysis patients without supplemental nutrition.

ELIGIBILITY:
Inclusion Criteria:

* patients on hemodialysis for more than 1 year,
* Group 1: HIV infection

Exclusion Criteria:

* patients on hemodialysis for less than 1 year,
* Group 2 and 3: HIV infection
* no pre-/post dialysis weight differences of > 3 kg after long HD free interval over last 10 HD sessions.
* no current high-caloric nutrition supplements or planned high-caloric supplements for clinical reasons.
* pregnancy
* for women: no use of oral contraceptives or other at least equally effective contraception in women with childbearing potential
* known neoplastic disease other than skin tumors (except melanoma)
* mental disease or retardation with impaired judgement power

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-09 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Cross sectional area of triceps m. in mid-humerus position (MRT) | 6 months

SECONDARY OUTCOMES:
plasma albumin < 3.6 mg/dl | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the Goethe University Frankfurt am Main, Frankfurt am Main, Germany

REFERENCES:
- [Derived] Zilles M, Betz C, Jung O, Gauer S, Hammerstingl R, Wachtershauser A, Vogl TJ, Geiger H, Asbe-Vollkopf A, Pliquett RU. How to Prevent Renal Cachexia? A Clinical Randomized Pilot Study Testing Oral Supplemental Nutrition in Hemodialysis Patients With and Without Human Immunodeficiency Virus Infection. J Ren Nutr. 2018 Jan;28(1):37-44. doi: 10.1053/j.jrn.2017.07.003. Epub 2017 Nov 14. PMID 29146139